CLINICAL TRIAL: NCT00358917
Title: A Phase 3, Randomized, Open-Label Study of Lopinavir/Ritonavir (LPV/r) Tablets 800/200 Milligram (mg) Once-Daily (QD) Versus 400/100 mg Twice-Daily (BID) When Coadministered With Nucleoside/Nucleotide Reverse Transcriptase Inhibitors (NRTIs) in Antiretroviral-Experienced, Human Immunodeficiency Virus Type 1 (HIV-1) Infected Subjects
Brief Title: Study of Lopinavir/Ritonavir Tablets Comparing Once-Daily Versus Twice-Daily Administration When Coadministered With Nucleoside/Nucleotide Reverse Transcriptase Inhibitors in Antiretroviral-Experienced Human Immunodeficiency Virus Type 1 Infected Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Barry Bernstein, MD, Project Director, Abbott
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M06-802
Record Dates: First submitted 2006-07-28; First posted 2006-08-01 (Estimated); Results first posted 2010-02-01 (Estimated); Last update posted 2011-04-11 (Estimated); Status verified 2011-04

CONDITIONS: Human Immunodeficiency Virus Infections
MeSH Terms: interventions — Lopinavir; Ritonavir; Tablets; lopinavir-ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LPV/r 800/200 mg QD Tablet (Experimental)
  Interventions: Drug: lopinavir/ritonavir (LPV/r) tablet with nucleoside/nucleotide reverse transcriptase inhibitors (NRTIs)
- LPV/r 400/100 mg BID Tablet (Active Comparator)
  Interventions: Drug: lopinavir/ritonavir (LPV/r) tablet with nucleoside/nucleotide reverse transcriptase inhibitors (NRTIs)

INTERVENTIONS:
Drug: lopinavir/ritonavir (LPV/r) tablet with nucleoside/nucleotide reverse transcriptase inhibitors (NRTIs) — LPV/r 800/200 mg once-daily (QD) tablet
  Other Names: ABT-378; lopinavir/ritonavir; Kaletra
  Arms: LPV/r 800/200 mg QD Tablet
Drug: lopinavir/ritonavir (LPV/r) tablet with nucleoside/nucleotide reverse transcriptase inhibitors (NRTIs) — LPV/r 400/100 mg twice-daily (BID) tablet
  Other Names: ABT-378; lopinavir/ritonavir; Kaletra
  Arms: LPV/r 400/100 mg BID Tablet

SUMMARY:
The purpose of this study was to compare the safety, tolerability, and antiviral activity of once-daily (QD) and twice-daily (BID) dosing of the lopinavir/ritonavir (LPV/r) tablet formulation in combination with nucleoside/nucleotide reverse transcriptase inhibitors (NRTIs) in antiretroviral-experienced human immunodeficiency virus type 1 infected subjects with detectable viral load while receiving their current antiretroviral therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects were human immunodeficiency virus type 1 (HIV-1) positive, antiretroviral-experienced adults at least 18 years of age currently receiving an antiretroviral regimen which had not changed for at least 12 weeks.
* Subjects had plasma HIV-1 ribonucleic acid (RNA) levels > 1,000 copies/mL at screening and were not acutely ill.
* Subject was currently failing his/her antiretroviral regimen with the most recent 2 consecutive prestudy plasma HIV-1 RNA levels > 400 copies/mL with the most recent being > 1000 copies/mL, and in the investigator's opinion, should change therapy
* Female subjects were nonpregnant and nonlactating.

Exclusion Criteria:

* Subjects were excluded if screening laboratory analyses showed hemoglobin <= 8.0 grams per deciliter.
* Subjects were excluded if screening laboratory analyses showed absolute neutrophil count <= 750 cells/microliter.
* Subjects were excluded if screening laboratory analyses showed platelet count <= 50,000 per cubic millimeter.
* Subjects were excluded if screening laboratory analyses showed alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >= 5.0 x upper limit of normal (ULN).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 599 (Actual)
Dates: Start 2006-08; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Podsadecki, MD, Study Director — Abbott
Locations (1):
- Medical Information - Abbott (1-800-633-9110), Abbott Park, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- LPV/r 800/200 mg QD Tablet: lopinavir/ritonavir 800/200 milligram (mg) once daily (QD) tablet
- LPV/r 400/100 mg BID Tablet: lopinavir/ritonavir 400/100 milligram (mg) twice daily (BID) tablet
Period: Overall Study
Arm/Group | LPV/r 800/200 mg QD Tablet | LPV/r 400/100 mg BID Tablet
Started | 300 | 299
Completed | 234 | 230
Not Completed | 66 | 69
Not completed — Adverse Event | 14 | 21
Not completed — Withdrawal by Subject | 5 | 7
Not completed — Lost to Follow-up | 20 | 17
Not completed — Noncompliance | 12 | 11
Not completed — Death | 2 | 3
Not completed — Virologic failure | 11 | 8
Not completed — Unable to Continue Participation | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- LPV/r 800/200 mg QD Tablet: lopinavir/ritonavir 800/200 mg once daily (QD) tablet
- LPV/r 400/100 mg BID Tablet: lopinavir/ritonavir 400/100 mg twice daily (BID) tablet
- Total: Total of all reporting groups
Arm/Group | LPV/r 800/200 mg QD Tablet | LPV/r 400/100 mg BID Tablet | Total
Number analyzed (Participants) | 300 | 299 | 599
Age Continuous [Mean (Standard Deviation); unit: years] | 40.4 (9.22) | 40.8 (8.63) | 40.6 (8.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 103 | 206
  Male | 197 | 196 | 393
Received Prior Nonnucleoside Reverse Transcriptase Inhibitor (NNRTI) [Number; unit: participants]
  Received Prior NNRTI | 264 | 241 | 505
  Did Not Receive Prior NNRTI | 36 | 58 | 94
Received Prior Nucleoside/nucleotide Reverse Transcriptase Inhibitor (NRTI) [Number; unit: participants]
  Received Prior NRTI | 299 | 297 | 596
  Did Not Receive Prior NRTI | 1 | 2 | 3
Received Prior Protease Inhibitor (PI) [Number; unit: participants]
  Received Prior PI | 140 | 136 | 276
  Did Not Receive Prior PI | 160 | 163 | 323
Cluster of Differentiation 4 Single-Positive Thymocyte (CD4+ T) Cell Count [Mean (Standard Deviation); unit: cells/microliter] | 239.3 (158.39) | 268.3 (183.55) | 253.9 (171.98)
Plasma Human Immunodeficiency Virus Type 1 (HIV-1) Ribonucleic Acid (RNA) Level [Mean (Standard Deviation); unit: log10 copies/milliliter (mL)] | 4.26 (0.826) | 4.26 (0.809) | 4.26 (0.817)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Responding at Week 48 Based on the Food and Drug Administration (FDA) Time to Loss of Virologic Response (TLOVR) Algorithm
Description: A participant was classified as a responder at the first of 2 consecutive human immunodeficiency virus type 1 (HIV-1) ribonucleic acid (RNA) levels <50 copies/mL. The participant continued to be a responder until 2 consecutive values >=50 copies/mL were reached, until the final value if that value was >=50 copies/mL, or until discontinuation or death.
Time Frame: Week 48 (End of Study)
Population: Intention to treat analysis of all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | LPV/r 800/200 mg QD Tablet | LPV/r 400/100 mg BID Tablet
Number analyzed (Participants) | 300 | 299
Percentage of Participants | 55.3 | 51.8
Statistical Analysis 1: Comparison: LPV/r 800/200 mg QD Tablet vs LPV/r 400/100 mg BID Tablet; The null hypothesis was that the response rate for the once daily (QD) regimen was more than 12% lower than the response rate for the twice daily (BID) regimen. The planned sample size of 600 participants (300 participants in each of the QD and BID treatment regimens) provided 83% power (with a type I error rate of 0.05) to reject the null hypothesis, i.e., to determine noninferiority based on the 12% margin; Test type: Non-Inferiority or Equivalence — The 95% confidence interval for the difference in response rates (once daily [QD] minus twice daily [BID], based on the normal approximation to the binomial distribution) was used to assess noninferiority. The QD regimen was considered noninferior to the BID regimen if the lower limit of the confidence interval remained above -12%; p = 0.413, normal approx. to binomial distribution; Diff. in Percentage of Subj. Responding = 3.5, 95% CI [-4.5 to 11.5]

2. Secondary Outcome: Percentage of Participants With Plasma Human Immunodeficiency Virus Type 1 (HIV-1) Ribonucleic Acid (RNA) Levels < 50 Copies/Milliliter (mL) at Week 48
Time Frame: Week 48 (End of Study)
Population: Observed data analysis using all available Week 48 data from all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | LPV/r 800/200 mg QD Tablet | LPV/r 400/100 mg BID Tablet
Number analyzed (Participants) | 225 | 223
Percentage of Participants | 76.0 | 72.2
Statistical Analysis 1: Comparison: LPV/r 800/200 mg QD Tablet vs LPV/r 400/100 mg BID Tablet; Test type: Superiority or Other; p = 0.389, normal approx. to binomial distribution; Diff. in Percentage of Subj. Responding = 3.8, 95% CI [-4.3 to 11.9]

3. Secondary Outcome: Mean Change From Baseline to Week 48 in Cluster of Differentiation 4 Single-Positive Thymocyte (CD4+ T) Cell Counts
Time Frame: Week 48 (End of Study)
Population: All randomized participants who received at least 1 dose of study drug and who had CD4+ T cell counts at both the Baseline Visit and Week 48.
Measure: Mean (Standard Error); unit: cells/microliter
Arm/Group | LPV/r 800/200 mg QD Tablet | LPV/r 400/100 mg BID Tablet
Number analyzed (Participants) | 195 | 193
cells/microliter | 135.3 (9.03) | 121.5 (9.08)
Statistical Analysis 1: Comparison: LPV/r 800/200 mg QD Tablet vs LPV/r 400/100 mg BID Tablet; Test type: Superiority or Other; p = 0.281, ANOVA

4. Secondary Outcome: Virologic Response (HIV-1 RNA <50 Copies/mL) at Week 48 for Participants With 0-2 Protease Inhibitor Substitutions at Baseline Associated With Reduced Response to Lopinavir/Ritonavir
Description: Substitutions considered in the analysis were L10F/I/R/V, K20M/N/R, L24I, L33F, M36I, I47V, G48V, I54L/T/V, V82A/C/F/S/T, and I84V as defined in the proposed United States Package Insert.
Time Frame: Week 48 (End of Study)
Population: Dropouts-as-censored: participants were responders if they had HIV-1 RNA <50 copies/mL at Week 48. Participants who discontinued (d/c'd) while suppressed or w/o post baseline (BL) levels were excluded. Those d/c'd <Day 85 were excluded unless they had >=1 post BL level & didn't achieve a decrease >=1.0 log10 copies/mL, then they were nonresponders.
Measure: Number; unit: Percentage of Participants
Groups:
- LPV/r 800/200 mg QD Tablet: lopinavir/ritonavir 800/200 mg once daily (QD) tablet; 88% NNRTI-experienced, 47% PI-experienced (24% nelfinavir, 19% indinavir, 13% atazanavir).
- LPV/r 400/100 mg BID Tablet: lopinavir/ritonavir 400/100 mg twice daily (BID) tablet; 81% NNRTI-experienced, 45% PI-experienced (20% nelfinavir, 17% indinavir, 13% atazanavir).
Arm/Group | LPV/r 800/200 mg QD Tablet | LPV/r 400/100 mg BID Tablet
Number analyzed (Participants) | 255 | 250
Percentage of Participants | 65.5 | 61.6

5. Secondary Outcome: Percentage of Participants With New Primary Protease Mutations at Week 48
Description: Emergence of new primary protease inhibitor mutations (i.e., mutations at codons 30, 32, 48, 50, 82, 84, and 90 that were not present at baseline).
Time Frame: Week 48 (End of Study)
Population: All randomized participants who received at least 1 dose of study drug and had post baseline genotypic resistance assay results.
Measure: Number; unit: Percentage of Participants
Arm/Group | LPV/r 800/200 mg QD Tablet | LPV/r 400/100 mg BID Tablet
Number analyzed (Participants) | 75 | 77
Percentage of Participants | 8.0 | 15.6
Statistical Analysis 1: Comparison: LPV/r 800/200 mg QD Tablet vs LPV/r 400/100 mg BID Tablet; Test type: Superiority or Other; p = 0.222, Fisher Exact

ADVERSE EVENTS:
Arm/Group | LPV/r 800/200 mg QD Tablet | LPV/r 400/100 mg BID Tablet
Serious Adverse Events (participants affected / at risk) | 27/300 | 37/299
Other Adverse Events (participants affected / at risk) | 201/300 | 180/299
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LPV/r 800/200 mg QD Tablet (N=300) | LPV/r 400/100 mg BID Tablet (N=299)
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 0
Tricuspid valve incompetence (Cardiac disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Asthenia (General disorders) | 0 | 1
Chest pain (General disorders) | 1 | 1
Chills (General disorders) | 1 | 0
Death (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 1
Unevaluable event (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1
Abscess limb (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Bacterial disease carrier (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Cerebral toxoplasmosis (Infections and infestations) | 1 | 0
Cryptococcosis (Infections and infestations) | 1 | 0
Dengue fever (Infections and infestations) | 1 | 0
Disseminated tuberculosis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Helicobacter infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 0 | 1
Meningitis tuberculous (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 3 | 5
Sepsis (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 1
Staphylococcal skin infection (Infections and infestations) | 0 | 1
Syphilis (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 0
Lung injury (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Scapula fracture (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0
Hyperlactacidaemia (Metabolism and nutrition disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Ocular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Encephalitis (Nervous system disorders) | 0 | 1
Mononeuritis (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 1
Major depression (Psychiatric disorders) | 1 | 0
Personality disorder (Psychiatric disorders) | 0 | 1
Acute prerenal failure (Renal and urinary disorders) | 1 | 0
Choluria (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1
Epididymitis (Reproductive system and breast disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1
Vaginal dysplasia (Reproductive system and breast disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4.9% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LPV/r 800/200 mg QD Tablet (N=300) | LPV/r 400/100 mg BID Tablet (N=299)
Abdominal pain (Gastrointestinal disorders) | 17 | 8
Diarrhoea (Gastrointestinal disorders) | 149 | 115
Nausea (Gastrointestinal disorders) | 47 | 66
Vomiting (Gastrointestinal disorders) | 36 | 37
Influenza (Infections and infestations) | 21 | 19
Nasopharyngitis (Infections and infestations) | 13 | 16
Upper respiratory tract infection (Infections and infestations) | 29 | 26
Headache (Nervous system disorders) | 20 | 21
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This study has varying agreements that have been negotiated individually; however, it appears that the most restrictive of the agreements states that following the first publication/presentation of the study by Abbott (or twelve [12] months after the completion of the study at all sites, whichever occurs first), the Principal Investigator (PI) shall, during a period of twelve (12) months, have the right to publish/present the results of the site.